CLINICAL TRIAL: NCT05668780
Title: Integrating Addiction and Infectious Diseases Services Into Primary Care in Rural Settings
Brief Title: Buprenorphine Integration Research and Community Health
Acronym: BIRCH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000034075; R01DA054703 (NIH)
Record Dates: First submitted 2022-12-19; First posted 2022-12-30 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder; HIV Infections; Hepatitis C
Keywords: Implementation Science; HIV; Medication for Opioid Use Disorder; PrEP; Hepatitis C; Nominal Group Technique
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections; Hepatitis C

STUDY DESIGN:
Intervention Model Description: Using a step-wedge design with 20 PCCs, the investigators will conduct a Type 3 Hybrid implementation trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention - Nominal Group Technique, Training, Coaching (Experimental): Each group of clinics will receive the same intervention in a step-wedge design, starting every 6-months.
  Interventions: Behavioral: NIATx Coaching

INTERVENTIONS:
Behavioral: NIATx Coaching — The intervention will consist of:
  1. a Nominal Group Technique session to identify priorities in integrating HIV/HCV/MOUD
  2. rapid cycle improvement coaching sessions from a NIATx coach, using data dashboards and screening alerts to improve identification and treatment for HIV/HCV/OUD
  3. training for primary care providers

SUMMARY:
The goal of this clinical trial is to evaluate an intervention strategy in introducing screen/evaluate/treat (SET) procedures for HIV/ hepatitis C/ and Opioid Use Disorder in Primary Care Clinics in West Virginia.

The main questions it aims to answer are:

* What are the barriers and facilitators to integrating evidence based practices for screening and treatment of HIV, hepatitis C, and Opioid Use Disorder into primary care clinics in West Virginia?
* To assess the extent to which our SET processes are achieved through enhanced EHR tools, NIATx (formerly known as Network for the Improvement of Addiction Treatment) facilitation and Extension for Community Healthcare Outcomes (ECHO)-supported collaborative learning?
* Does implementing these services improve primary and secondary health outcomes for patients? Primary Care Clinics will participate in training and process improvement coaching to integrate these services. Using a step-wise design, 20 Primary Care Clinics will undergo the training and coaching in four groups of five clinics.

DETAILED DESCRIPTION:
To integrate HIV/HCV/ OUD services into Primary Care Clinics (PCC), the investigators will introduce screen/evaluate/treat (SET) procedures for HIV/hepatitis C (HCV)/ Opioid Use Disorder (OUD) in PCCs in rural WV where ECHO and WV Hepatitis Academic Mentoring Partnership (WVHAMP) will support clinical skills for Primary Care Provider (PCPs) and where NIATx process improvement tools will be used to guide adoption and scale-up of SET procedures to achieve integration. Using a step-wedge design with 20 PCCs, the investigators will conduct a Type 3 Hybrid implementation trial and examine the extent to which our SET processes are achieved through enhanced electronic health record (EHR) tools, NIATx facilitation and ECHO and WVHAMP collaborative learning. Implementation outcomes include adoption of screening and treating with three distinct but linked evidence based practices (EBPs) for OUD, HIV and HCV in PCCs. Effectiveness outcomes will include quality health indicators (QHIs) for primary care, HIV, HCV and OUD.

This project is separated into two Phases. Phase 1 includes Nominal Group Technique focus groups and anonymous staff surveys at the 20 PCCs to identify barriers and facilitators to integrating these evidence based practices. Phase 2 is an evaluation of deidentified reports from the PCCs Electronic Health Records. In Phase 2, randomized sites will start NIATx activities, including a series of rapid-cycle Plan-Do-Study-Act (PDSA) activities. The first 6 months will include intensive coaching from a certified NIATx coach and enhanced by support from ECHO & the WVHAMP to teach subspecialty clinical expertise. During an 18-month follow-up, the investigators will assess the sustainability of these practice changes. Effectiveness outcomes will include a set of nationally recommended quality health indicators (QHIs) to measure quality care. This project is a collaboration between Yale University, West Virginia University (WVU), and the West Virginia Primary Care Association.

Aim 1 (Phase 1):

Identify the barriers and facilitators for a diverse group of PCCs throughout WV, a mostly rural state that is profoundly impacted by OUD-associated HIV/HCV outbreaks, focusing on screening for and prescribing evidence-based treatment [medication for opioid use disorder (MOUD), Treatment as Prevention (TasP), pre-exposure prophylaxis (PrEP), and curative hepatitis C (HCV) treatment] for OUD, HIV and HCV.

Aim 2 (Phase 2):

Using a step-wedge design with 20 PCCs, the investigators will conduct a Type 3 hybrid implementation trial using the Integrated Promoting Action on Research Implementation in Health Services (iPARiHS) framework to assess the extent to which our SET processes are achieved through enhanced EHR tools, NIATx facilitation and ECHO-supported collaborative learning. Implementation outcomes include adoption of screening and implementation of three distinct but linked EBPs for OUD, HIV and HCV in PCCs. Effectiveness outcomes will include quality health indicators (QHIs) for primary care, HIV, HCV and OUD.

ELIGIBILITY:
Inclusion Criteria:

- Federally Qualified Health Centers (FQHCs) and Look-Alike FQHC Primary Care Clinics in West Virginia providing adult care

Exclusion Criteria:

* Clinics (private or specialty) or any clinics not in West Virginia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Organizational Readiness and Staff Attitudes towards integration of OUD, HIV, HCV services into primary care clinics | Every 6 months for 24 months
  Staff survey results on organizational capacity, readiness to change, organizational functioning and social dominance orientation, and resistance to change.
Integration of services | 24 months
  Adoption of screening and implementation of best evidence-based practices. Quality health indicators (QHIs) for primary care - OUD, HIV & HCV documented in electronic health record data.
Number of patients screened for opioid use disorder (OUD) | 18 months
  Screening result for opioid use disorder documented in electronic health record (EHR)
Number of patients initiated on medications for OUD | 18 months
  Prescription medication for OUD; prescription dates, medication type
Number of patients screened for HIV | 18 months
  Lab ordered and result for HIV test entered in EHR
Number of patients initiated on antiretroviral medication (ART) for HIV | 18 months
  For those with a positive HIV test result, prescription medication for HIV; prescription dates
Number of patients screened for Hepatitis C (HCV) | 18 months
  Lab result ordered for HCV antibody / reflex polymerase chain reaction (PCR), result entered in EHR
Number of patients initiated on medication for HCV | 18 months
  For those with a positive HCV PCR test, documented in EHR prescription medication for HCV; prescription dates; fibrosis score
Number of patients prescribed PrEP | 18 months
  For those with a negative HIV result, prescription medication for PrEP; medication type; prescription dates; lab orders

SECONDARY OUTCOMES:
Number of patients with sustained viral response for HCV | 18 months
  For those with HCV medication prescription; Viral load results in EHR after recommended treatment
Number of patients retained on medication for OUD for at least 6 months | 6 months
  For those with prescription for medication for OUD; documentation in EHR of repeated prescription orders
Number of patients retained on medication (ART) for HIV | 12 months
  For those with new prescription for medication for HIV; documentation in EHR of repeated prescriptions up to 6 and 12 months
Number of patients with Viral Suppression for HIV | 12 months
  For those with new HIV diagnosis; documentation in EHR of viral suppression defined as HIV RNA <200 copies/µl, at 6 and 12 months after prescription
Number of patients on PrEP to prevent HIV | 12 months
  Documentation of negative HIV labs in EHR every 3 months
Quality Health Indicator (QHI) score for Primary Care screening variables | 18 months
  QHI-PC score based on documentation of screening (limited age/sex) for hypertension, diabetes, hyperlipidemia, HIV, HCV, hepatitis B (HBV), syphilis, cervical cancer, breast cancers, prostate cancer, herpes simplex virus (HSV) serology, latent tuberculosis (TB), colorectal cancer, depression, chlamydia, gonorrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Yale University; Natalie Kil, MPH, Study Director — Yale University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No